CLINICAL TRIAL: NCT06745804
Title: Phase 1 Imaging Study of 68Ga-R10602-101 in Hormone Receptor-Positive Breast Cancer
Brief Title: Study of 68Ga-R10602
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Radionetics Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: R10602-101
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-07

CONDITIONS: Locoregionally Recurrent Hormone-receptor Positive Breast Cancer; Metastatic Hormone Receptor Positive Breast Cancer; Hormone Receptor Positive Breast Adenocarcinoma
Keywords: Hormone Receptor Positive Breast Cancer; Endocrine resistant; Radioisotope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 68Ga-R10602 Imaging Optimization Portion (Cohort 1) (Other): 68Ga-R10602 injection at pre-defined dose levels. PET/CT imaging at pre-defined timepoints.
  Interventions: Drug: 68Ga-R10602 injection
- 68Ga-R10602 Imaging Confirmation Portion (Cohort 2) (Other): 68Ga-R10602 injection at the selected dose level. PET/CT imaging at a single timepoint.
  Interventions: Drug: 68Ga-R10602 injection

INTERVENTIONS:
Drug: 68Ga-R10602 injection — 68Ga-R10602 is a gallium-labeled small molecule radioligand that is designed to localize tumor lesions in hormone receptor positive breast cancer

SUMMARY:
A phase 1 imaging study of 68Ga-R10602 in hormone-receptor positive breast cancer.

DETAILED DESCRIPTION:
There are three eligible disease populations for the study. Population 1 are patients with metastatic or locoregionally recurrent, endocrine-resistant, ER+ and/or PR+ breast cancer who have received at least one line of chemotherapy or ADC. Population 2 are patients with ER+ and HER2- locoregional or metastatic non-resectable breast adenocarcinoma with progression on at least one line of prior endocrine therapy in the adjuvant or metastatic setting and starting next line of therapy that will include tamoxifen, fulvestrant, aromatase inhibitor, or elacestrant with or without ovarian suppression. Population 3 are patients with ER+ and/or PR+ and HER2- breast cancer who are ineligible for Population 1 or 2. All disease populations are eligible for both cohorts.

Cohort 1 will consist of three dose de-escalating cohorts with four patients each for a total of twelve patients. Once the twelve patients have completed the dose de-escalation, the three dose levels will be evaluated, and additional subjects may be enrolled into Cohort 1 at the single chosen dose. All patients will undergo imaging at a single timepoint and no dosimetry will be performed.

In Cohort 2, approximately six to eight patients will receive the single chosen dose followed by imaging at five timepoints and blood dosimetry at seven timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Breast Cancer Eligibility:

   * Population 1: Pathologically confirmed ER and/or PR positive, locoregionally recurrent or metastatic breast cancer that is refractory to endocrine therapy (progression on at least one line of endocrine therapy and determined by the investigator that Study Participant would not benefit from additional endocrine therapy) who have received at least one line of chemotherapy or antibody drug conjugate in the metastatic setting (recurrence within 6 months of adjuvant chemotherapy counts as one line of therapy). There is no limit on prior number of lines of endocrine therapy. Prior treatment with CDK4/6, AKT, PI3K and/or mTOR inhibitors is permitted.
   * Population 2: Pathologically confirmed ER positive and HER2 negative locoregional or metastatic breast adenocarcinoma that is not amenable to resection, with progression on at least one line of prior endocrine therapy in the adjuvant or metastatic setting and starting next line of therapy that will include endocrine therapy, such as tamoxifen, fulvestrant, aromatase inhibitor, or elacestrant with or without ovarian suppression.
   * Population 3: Study Participants with pathologically confirmed, estrogen and/or progesterone receptor (ER and/or PR) positive and HER2 negative breast adenocarcinoma who are ineligible for Population 1 or 2.
2. At least one target or non-target lesion per RECIST 1.1
3. Male or non-pregnant, non-lactating female Study Participant age ≥18 years. Female Study Participant of child-bearing potential and male Study Participant (if sexually active) must agree to use adequate method(s) of effective contraception during their participation in the study.

   1. Medically acceptable adequate contraception for sexually active females with child-bearing potential include: 1) surgical sterilization (such as tubal ligation or hysterectomy), 2) approved hormonal contraceptives, 3) barrier method (such as condom or diaphragm) used with a spermicide, or 4) intrauterine device (IUD).
   2. Medically acceptable adequate contraception for sexually active males include: 1) surgical sterilization (such as vasectomy), 2) a condom used with a spermicide.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
5. Adequate hepatic function as defined below (within 28 days of dosing with 68Ga R10602):

   1. Serum alanine aminotransaminase (ALT)/ aspartate aminotransaminase (AST) ≤3 × upper limit of normal (ULN) or ≤5 × ULN if liver metastases are present, and
   2. Serum bilirubin: total ≤1.5 × ULN (unless due to Gilbert's syndrome or hemolysis in which case total ≤3.0 × ULN).
6. Adequate renal function as measured by creatinine clearance calculated by the Cockcroft-Gault formula (≥60 mL/minute), determined within 28 days of dosing with 68Ga-R10602.
7. Able to understand and willing to sign an informed consent form (ICF).

Exclusion Criteria:

1. Received a radionuclide within a period of less than 10 physical half-lives of the administered radionuclide prior to dosing with 68Ga-R10602.
2. Radiotherapy ≤14 days prior to dosing with 68Ga-R10602.
3. Major surgery ≤21 days prior to dosing with 68Ga-R10602 or has not recovered from adverse effects of such procedure.
4. Severe or unstable medical condition, such as congestive heart failure (New York Heart Association [NYHA] Class III or IV), ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, as well as an uncontrolled cardiac arrhythmia requiring medication (≥Grade 2, according to NCI-CTCAE Version 5.0), myocardial infarction within 6 months prior to starting Investigational Product, or any other significant or unstable concurrent cardiac illness. Note: Stable chronic atrial fibrillation is allowed.
5. History of cerebrovascular accident within 6 months or that resulted in ongoing neurologic instability.
6. Major active infection requiring antibiotics.
7. Known active human immunodeficiency virus infection or active infection with Hepatitis B or C.
8. Acute illness within 14 days prior to dosing with 68Ga-R10602 unless mild in severity, as assessed by the Investigator.
9. Any other condition that in the opinion of the Investigator would place the Study Participant at an unacceptable risk or cause the Study Participant to be unlikely to fully participate or comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Day 1 to Day 7
  Number of participants with adverse events as assessed by NCI-CTCAE v5.0, including grade
Incidence of Serious Adverse Events | Day 1 to Day 7
  Number of participants with serious adverse events
Incidence of Clinically Significant Lab Changes | Day 1 to Day 7
  Number of participants with clinically significant change in clinical laboratory parameters

SECONDARY OUTCOMES:
Number and location of tumors identified by 68Ga-R10602 PET/CT | 1 day
  Number of tumors identified by 68Ga-PET/CT per participant
Number and location of tumors identified by 68Ga-R10602 PET/CT | 1 Day
  Location of tumors identified by 68Ga-10602 PET/CT per participants
Number and location of tumors identified by 68Ga-R10602 PET/CT | 1 Day
  SUV max of tumor lesions per participant
Number and location of tumors identified by 68Ga-R10602 PET/CT | 1 Day
  Ratio of tumor SUV over reference regions SUV
Number and location of tumor lesions identified by 68Ga-R10602 PET/CT versus standard of care imaging | 1 day
  Number and location of tumor lesions identified by 68Ga-R10602 PET/CT and by standard of care imaging (e.g. contrast enhanced diagnostic CT) and concordance rate between 68Ga-R10602 PET/CT and standard of care images.
Image quality | 1 day
  Image quality as assessed by a 5-point Likert scale by central review
Absorbed dose coefficients and total body effective dose | 1 day
  Absorbed dose coefficients (milliGray [mGy]/megabecquerel [MBq]) in organs.
Absorbed dose coefficients and total body effective dose | 1 Day
  The total body effective dose (milliSievert [mSv]/MBq).
PK parameters | 1 day
  PK parameters, including Cmax
PK parameters | 1 Day
  PK parameters including area under the curve (AUC).
PK parameters | 1 Day
  PK parameters including half-life (T1/2) in blood samples.
PK parameters | 1 Day
  Other pharmacokinetic (PK) parameters may also be evaluated as needed to support the outcome measure.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Michigan Medicine, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No